CLINICAL TRIAL: NCT01405872
Title: An Observational Study to Assess Persistence, Adherence, Quality of Life, and Treatment Satisfaction in Patients Beginning Therapy With the Avonex® PEN™.
Brief Title: Persistence, Adherence, Quality of Life, and Treatment Satisfaction With Avonex® PEN™.
Acronym: PERSIST
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 108MS402
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: AVONEX PEN — Participants receive Avonex PEN commercially prescribed according to the local prescribing information.

SUMMARY:
The primary objective of the study is to determine physician reported persistence with the Avonex PEN at Month 12/End of Study as well as determining factors associated with persistence. The secondary objectives for this study are as follows: To evaluate the tolerability for treatment administration of the Avonex PEN at Months 3, 6, and 12; To evaluate patient quality of life (QoL) while using the Avonex PEN for treatment administration at Months 3, 6, and 12; To evaluate clarity of directions for use of the Avonex PEN at Month 3; To evaluate ease of use and the patient's assessment of the injection procedure with the Avonex PEN at Months 3, 6, and 12; To evaluate patient reported adherence at Months 6 and 12; To evaluate physician reported persistence at Month 6; To evaluate overall patient satisfaction with the use of the Avonex PEN for treatment administration at Months 3, 6, and 12; To evaluate patient reported fear of injection at Months 3, 6, and 12; and To evaluate the percentage of patients switching from caregiver to self-injection at Months 3, 6, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent
* Must satisfy the locally approved therapeutic indications for the Avonex PEN
* Decision to treat with Avonex PEN must precede enrollment
* Must have no more than two (2) injections with the Avonex PEN prior to enrollment

Exclusion Criteria:

* Inability to comply with study requirements
* Other unspecified reasons that, in the opinion of the investigator or Biogen Idec, make the patient unsuitable for enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Multiple Sclerosis patients who have made the decision, along with their health care provider, to begin therapy with Avonex PEN.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Persistence with Avonex PEN therapy at Month 12/End of Study as measured by the percentage of patients remaining on therapy at Month 12/End of Study as reported by a physician. | 12 months

SECONDARY OUTCOMES:
Tolerability of Avonex PEN as measured by Injection Site Pain | Months 3, 6, and 12
Patient Quality of Life as measured by the EuroQol 5 domain (EQ-5D) Questionnaire | Months 3, 6, and 12
Clarity of directions for use of the Avonex PEN as measured by the Avonex PEN Instruction Grading Scale | Month 3
Ease of use and patient's assessment of the injection procedure with the Avonex PEN as measured by Ease of Use Grading Scale | Months 3, 6, and 12
Patient reported adherence as measured by number of doses missed | Over the first 6 months and during Months 6 & 12
Physician reported persistence as measured by number of patients still on therapy | Month 6
Patient reported satisfaction with the Avonex PEN as measured by the Patient Satisfaction Questionnaire | Months 3, 6 and 12
Patient reported fear of injection using the Fear of Injection Scale | Months 3, 6 and 12
Percent of patients switching from caregiver to self-injection | Months 3, 6, and 12
Tolerability of Avonex PEN as measured by Injection Site Reaction | Months 3, 6 and 12
Ease of use and patient's assessment of the injection procedure with the Avonex PEN as measured by Patient Assessment of Injection Procedure | Months 3, 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (64):
- Denmark (3):
  - Research Site, Glostrup Municipality
  - Research Site, Holstebro
  - Research Site, Næstved
- France (6):
  - Research Site, Amiens
  - Research Site, Clermont-Ferrand
  - Research Site, Créteil
  - Research Site, Nancy
  - Research Site, Rouen
  - Research Site, Strasbourg
- Germany (25):
  - Research Site, Aachen
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Eisenach
  - Research Site, Erbach im Odenwald
  - Research Site, Freiburg im Breisgau
  - Research Site, Hamburg
  - Research Site, Heidenheim
  - Research Site, Herford
  - Research Site, Itzehoe
  - Research Site, Kastellaun
  - Research Site, München
  - Research Site, Nagold
  - Research Site, Potsdam
  - Research Site, Regensburg
  - Research Site, Rottweil
  - Research Site, Rüdersdorf
  - Research Site, Schwendi
  - Research Site, Siegen
  - Research Site, Sinsheim
  - Research Site, Stade
  - Research Site, Weil am Rhein
  - Research Site, Weisbaden
  - Research Site, Wolfratshausen
- Netherlands (5):
  - Research Site, 's-Hertogenbosch
  - Research Site, Eindhoven
  - Research Site, Heerlen
  - Research Site, Leeuwarden
  - Research Site, Sittard
- Norway (5):
  - Research Site, Bergen
  - Research Site, Drammem
  - Research Site, Førde
  - Research Site, Molde
  - Research Site, Tønsberg
- Research Site, Amadora, Portugal
- Research Site, Košice, Slovakia
- Sweden (7):
  - Research Site, Helsingborg
  - Research Site, Karlstad
  - Research Site, Linköping
  - Research Site, Norrköping
  - Research Site, Skövde
  - Research Site, Stockholm
  - Research Site, Trollhättan
- Switzerland (4):
  - Research Site, Lucerne
  - Research Site, Lugano
  - Research Site, Sankt Gallen
  - Research Site, Sion
- United Kingdom (7):
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Hammersmith
  - Research Site, Haywards Heath
  - Research Site, Irvine
  - Research Site, Leicester
  - Research Site, Sheffield

REFERENCES:
- [Derived] Hupperts R, Becker V, Friedrich J, Gobbi C, Salgado AV, Sperling B, You X. Multiple sclerosis patients treated with intramuscular IFN-beta-1a autoinjector in a real-world setting: prospective evaluation of treatment persistence, adherence, quality of life and satisfaction. Expert Opin Drug Deliv. 2015 Jan;12(1):15-25. doi: 10.1517/17425247.2015.989209. Epub 2014 Nov 28. PMID 25430947